CLINICAL TRIAL: NCT04373980
Title: Conventional Versus LED Phototherapy and Their Effect on Lymphocytes Subsets of Full Term Neonates With Hyperbilirubinemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rania Ali El-Farrash (Other)
Responsible Party: Sponsor-Investigator, Rania Ali El-Farrash, Assistant professor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: FMASU 000017585
Record Dates: First submitted 2020-04-28; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Neonatal Hyperbilirubinemia; Phototherapy Complication
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal | interventions — Phototherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional phototherapy (Active Comparator): neonates with unconjugated hyperbilirubinemia exposed to conventional phototherapy
  Interventions: Device: phototherapy
- LED phototherapy (Active Comparator): neonates with unconjugated hyperbilirubinemia exposed to LED phototherapy
  Interventions: Device: phototherapy
- Control group (No Intervention)

INTERVENTIONS:
Device: phototherapy — estimate CD4 and CD8 subsets in neonates with unconjugated hyperbilirubinemia after exposure to phototherapy
  Arms: LED phototherapy; conventional phototherapy

SUMMARY:
The aim of this study is to investigate the influence of the use of different types of phototherapy on different lymphocytes subsets CD4 and CD8 in the treatment of hyperbilirubinemia in neonates.

ELIGIBILITY:
Inclusion Criteria:

Term neonates with a gestational week higher than 37weeks, according to the guidelines of the American Academy of Pediatrics (2004) which stated that gestational ages of newborns are determined according to the first day of the mother's last menstrual period (by the mother's statement) and were additionally confirmed by the Ballard scoring system (Ballard et al., 1991) and antenatal ultrasonographic estimation or obstetric records if present.

* Clinically significant indirect hyperbilirubinemia requiring phototherapy in the first week of life.
* No pathologic etiological factors for hyperbilirubinemia

Exclusion Criteria:

* Total bilirubin level of >20 mg/dl.
* Prematurity.
* Sepsis.
* Congenital anomaly.
* Elevation in direct bilirubin level.
* History of immune deficiency the family.
* History of preeclampsia or any other diseases or drug use of the mother

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Effect of types of phototherapy on change in CD4 and CD8 lymphocytes subsets | 2 days
  Detection of CD4 and CD8 absolute counts(x10³/uL) : was done before and 48 hours after phototherapy and for controls at time of examination using monoclonal antibodies and measured by flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt